CLINICAL TRIAL: NCT05064943
Title: Reliability and Validity of the 2-Minute Step Test in Patients With Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hakan AKKAN, Assistant professor (Principal Investigator), Kutahya Health Sciences University
Other Study IDs: KutahyaHSU-AKKAN001
Record Dates: First submitted 2021-09-04; First posted 2021-10-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Total Knee Replacement; Reliability and Validity
Keywords: Total Knee Replacement; Step Test
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Knee Replacement: Patients who have undergone total knee replacement
  Interventions: Diagnostic Test: 2-minute step test

INTERVENTIONS:
Diagnostic Test: 2-minute step test — The participant stands and counts for 2 minutes. The minimum height to raise the knee is determined for each participant by calculating the midpoint between the patella and the anterior superior iliac spine. They are instructed to complete as many steps as possible during the 2-minute period. A verbal command is given every 30 seconds to encourage performance: "You're doing great, keep it up." If the claudication symptom becomes unbearable, the patient can stop during the test, but the time is not stopped. Patients who discontinue testing due to symptoms of claudication are encouraged to return to testing as soon as possible. An evaluator records the number of steps in the right leg.

SUMMARY:
Total knee arthroplasty (TKA) is a cost-effective treatment for end-stage knee osteoarthritis. It has demonstrable benefits such as reducing pain and improving activity and quality of life. Despite the decrease in pain after surgery, the expectations of patients regarding their physical functions are not fully realized. Physical performance tests and reporting tests are used to objectively evaluate physical function and reveal the patient's condition. It is known that physical performance tests better reflect post-surgical changes. In addition, it has been stated that there may be serious differences between the results of the reports based tests and the actual functional capacities of the patients. The 2-minute walk test and the 6-minute walk test are tests that are used in the evaluation of lower extremity physical performance and have been shown to be valid and reliable in different populations. However, a certain length of corridor is needed in order to carry out these timed walking tests. As an alternative to these, another test used in the evaluation of physical performance is the 2-minute step test. This test, which was developed in 1999, does not require much equipment and space, so the test can be easily applied in any environment. In this test, a height specific to each individual is determined (as high from the ground as the distance between the Spina iliaca anterior superior and the midpoint of the patella), and the participant is asked to raise and lower both knees, respectively, to this height for 2 minutes. These tests used in the evaluation of patients should be valid, reliable and sensitive. In clinical studies, reliability is an important psychometric property. Because stable data are necessary to provide accurate data on treatment effects or the amount of change observed over time. Another important psychometric property is validity. Validity is defined as the degree to which a concept is accurately measured in a quantitative study. Reliability studies of the 2-minute step test in active and sedentary lean adults have been conducted, but the psychometric evaluations necessary for its routine use in patients with TDP have not been performed.

DETAILED DESCRIPTION:
This study is a non-experimental, descriptive methodological study. Forty-nine patients who applied to the outpatient clinic of Kütahya Health Sciences University, Evliya Çelebi Training and Research Hospital due to knee osteoarthritis, will included in the study. Pre-study power analysis was performed and the power to detect clinically significant difference was calculated as 90% (5% Type I error level). The smallest sample size to be taken was determined by using the sample size creation section in the G-Power (version 3.0.10) program.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having been diagnosed with knee OA by an orthopedic specialist and having a knee prosthesis applied.

Exclusion Criteria:

* Those who do not understand verbal and written information in Turkish
* Patients who underwent complex surgery requiring bone grafting
* Those with orthopedic or neurological disease causing gait disturbance
* Those with pain of 5 or more on the numerical pain scale
* Those with a history of Myocardial Infarction
* Those who have undergone surgery in the last 6 months
* Those with concomitant heart failure
* Those with unstable angina
* Those with uncontrolled hypertension
* Those with severe COPD, Asthma and Interstitial Lung Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone total knee replacement surgery with age of older than 18.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Hospital for Special Surgery Knee-Rating Scale | Baseline
  The Hospital for Special Surgery knee-rating scale was developed to be used as a standardized tool to measure outcomes in patients with osteoarthritis and knee arthroplasty. The scale can be used to evaluate the patient before surgery and to monitor knee function after surgery. Hospital for Special Surgery knee rating scale is widely used in the clinic by physiotherapists and orthopaedic surgeons.
Numerical Pain Scale | Baseline
  The pain levels of the patients will be determined using the Numerical Pain Scale (NPS). This scale is a score containing values between 0-10 on a 10 cm horizontal line. In scoring, 0 points indicates the absence of pain, while 10 points means unbearable pain. Patients are asked to mark the part that is equivalent to their own pain on the 10 cm line. Thus, the pain level of the patients is determined.
2-Minute Step Test | Baseline
  The participant stands and counts for 2 minutes. The minimum height to raise the knee is determined for each participant by calculating the midpoint between the patella and the anterior superior iliac spine. They are instructed to complete as many steps as possible during the 2-minute period. A verbal command is given every 30 seconds to encourage performance: "You're doing great, keep it up." If the claudication symptom becomes unbearable, the patient can stop during the test, but the time is not stopped. Patients who discontinue testing due to symptoms of claudication are encouraged to return to testing as soon as possible. An evaluator records the number of steps in the right leg.
6-Minute Walking Test | Baseline
  The participant is asked to walk as far as possible along a 30-meter straight corridor in a 6-minute period. Running is not allowed. The evaluator gives the standard incentive "you are doing well, keep going" every minute during the test. The distance traveled in 6 minutes is recorded in meters.
2-Minute Walk Test | Baseline
  Participants are asked to walk within 2 minutes along a 30 m indoor corridor. They are not allowed to talk while walking. The distance walked is recorded in meters.
2-Minute Step Test | Within same day after the baseline
  The participant stands and counts for 2 minutes. The minimum height to raise the knee is determined for each participant by calculating the midpoint between the patella and the anterior superior iliac spine. They are instructed to complete as many steps as possible during the 2-minute period. A verbal command is given every 30 seconds to encourage performance: "You're doing great, keep it up." If the claudication symptom becomes unbearable, the patient can stop during the test, but the time is not stopped. Patients who discontinue testing due to symptoms of claudication are encouraged to return to testing as soon as possible. An evaluator records the number of steps in the right leg.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Akkan, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nogueira MA, Almeida TDN, Andrade GS, Ribeiro AS, Rego AS, Dias RDS, Ferreira PR, Penha LRLN, Pires FO, Dibai-Filho AV, Bassi-Dibai D. Reliability and Accuracy of 2-Minute Step Test in Active and Sedentary Lean Adults. J Manipulative Physiol Ther. 2021 Feb;44(2):120-127. doi: 10.1016/j.jmpt.2020.07.013. Epub 2021 Jan 9. PMID 33431278
- [Background] Ricci PA, Cabiddu R, Jurgensen SP, Andre LD, Oliveira CR, Di Thommazo-Luporini L, Ortega FP, Borghi-Silva A. Validation of the two-minute step test in obese with comorbibities and morbidly obese patients. Braz J Med Biol Res. 2019;52(9):e8402. doi: 10.1590/1414-431X20198402. Epub 2019 Aug 29. PMID 31482976
- [Background] Braghieri HA, Kanegusuku H, Corso SD, Cucato GG, Monteiro F, Wolosker N, Correia MA, Ritti-Dias RM. Validity and reliability of 2-min step test in patients with symptomatic peripheral artery disease. J Vasc Nurs. 2021 Jun;39(2):33-38. doi: 10.1016/j.jvn.2021.02.004. Epub 2021 Mar 19. PMID 34120695
- [Result] Akkan H, Kaya Mutlu E, Kuyubasi SN. Reliability and validity of the two-minute step test in patients with total knee arthroplasty. Disabil Rehabil. 2024 Jul;46(14):3128-3132. doi: 10.1080/09638288.2023.2239141. Epub 2023 Jul 24. PMID 37486184